CLINICAL TRIAL: NCT02198963
Title: Phase 1 21-Day Evaluation of the Cumulative Irritation Potential of RUT058-60 on Abraded and Non-Abraded Skin Sites
Brief Title: 21 Day Cumulative Skin Irritation of RUT058-60
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP01-117838; 130932-304.01 (Other: BioScience Laboratories, Inc)
Record Dates: First submitted 2014-07-18; First posted 2014-07-24 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Irritation/Irritant
Keywords: Skin irritation potential of RUT058-60.
MeSH Terms: interventions — Sodium Dodecyl Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hypochlorous acid Solution 106 mg/L (Experimental): Occlusive patches will be used to apply approximately 0.02 mL of the Test Product RUT058-60 to abraded and non-abraded sites on the skin in the scapular region of each subject's back.
  Interventions: Drug: Hypochlorous acid solution 106 mg/L
- 0.1% (w/v) Sodium Lauryl Sulfate (Active Comparator): Occlusive patches will be used to apply approximately 0.02 mL of the Positive Control (0.1% Sodium Lauryl Sulfate) to abraded and non-abraded sites on the skin in the scapular region of each subject's back, once daily for 21 days.
  Interventions: Drug: 0.1% (w/v) Sodium Lauryl Sulfate
- 0.9% Physiological Saline, USP (Placebo Comparator): Occlusive patches will be used to apply approximately 0.02 mL of the Negative Control (0.9% Physiological Saline, USP) to abraded and non-abraded sites on the skin in the scapular region of each subject's back, once daily for 21 days.
  Interventions: Drug: 0.9% Physiological Saline, USP

INTERVENTIONS:
Drug: Hypochlorous acid solution 106 mg/L — test product
  Other Names: RUT058-60
  Arms: Hypochlorous acid Solution 106 mg/L
Drug: 0.1% (w/v) Sodium Lauryl Sulfate — positive control
  Other Names: SLS
  Arms: 0.1% (w/v) Sodium Lauryl Sulfate
Drug: 0.9% Physiological Saline, USP — negative control
  Other Names: sterile saline
  Arms: 0.9% Physiological Saline, USP

SUMMARY:
The purpose of this study is to determine the skin irritation potential of RUT058-60 after repetitive patch application to abraded and non-abraded skin of human subjects.

DETAILED DESCRIPTION:
This Cumulative Irritation Evaluation is designed to determine the skin irritation potential of RUT058-60, after repetitive patch application to abraded and non-abraded skin of healthy human subjects. Abraded skin will be challenged because the Test Product may be used, in practice, on non-intact skin. The primary research objective in this study is determine the skin irritation potential of RUT058-60. This question will be answered based on the observed results acquired evaluating its application to the abraded and non-abraded skin of at least 30 volunteer subjects, on the test product relative to the control readings.

A sufficient number of subjects will be recruited into the study to ensure 30 subjects, including both males and females, complete the study. Prior to the first application of test materials, designated skin sites will be abraded using the Tape Stripping Procedure. Occlusive patches will be used to apply approximately 0.02 mL of Test Product, Positive Control and Negative Control to abraded and non-abraded sites on the skin in the scapular region of each subject's back. The irritation potential of the test materials will be determined over the course of a 21-day challenge period on at least 30 subjects. A test material will be applied to the same site, abraded and non-abraded, on each day for 21 days. The six skin sites will be evaluated visually prior to each patch application and following the final patch removal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be of either sex, at least 18 years of age and of any race
* Subjects must be free of tattoos, sunburn, dermatoses, cuts, lesions, or other disorders on the parascapular skin of the back
* Subjects must be in good general health, as evidenced by the Subject Confidential Information and Acceptance Criteria and confirmed by screening laboratory evaluations
* Subjects must read and sign an Informed Consent Form, Subject Confidential Information and Acceptance Criteria, Authorization to Use and Disclose Protected Health Information Form

Exclusion Criteria:

* Known allergies to latex (rubber), metals, ink, tape and/or adhesives, soap, hypochlorous acid, sodium lauryl sulfate, physiological Saline
* Exposure of the upper back region to antimicrobial agents, medicated soaps, medicated shampoos, medicated lotions, or strong detergents in the 7 days prior to, or during the 3-week test period; or sun-tanning, use of tanning beds, or swimming or soaking in pools or hot tubs
* Use of topical or systemic corticosteroid, antihistamine, or anti-inflammatory medications in the 7 days prior to, or during the 3-week test period
* A medical diagnosis of a physical condition, such as a current or recent severe illness, asthma, diabetes, hepatitis, an organ transplant, mitral valve prolapse, congenital heart disease, internal prostheses, or any immunocompromised condition, such as AIDS (or HIV positive)
* Pregnancy, plans to become pregnant within the pre-test period or test days of the study, or nursing a child. Women cannot be pregnant, as evidenced by a negative urine pregnancy test, or should be of non-childbearing potential; that is, surgically sterile or postmenopausal (amenorrhea for at least 12 months)
* Any active skin rashes or breaks in the skin of the parascapular region of the back
* Any sunburn or tattoos on the skin of the parascapular region of the back
* A currently active skin disease or inflammatory skin condition, including contact dermatitis
* Participation in a clinical study in the past 7 days or current participation in another clinical study
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator, should preclude participation
* Clinical laboratory assessments that are determined by the Principal Investigator to indicate a clinically relevant abnormality and/or an exclusionary medical condition
* Unwillingness to fulfill the performance requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pullman, M.D., Principal Investigator — BioScience Laboratories, Inc.
Locations (1):
- BioScience Laboratories, Inc., Butte, Montana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and screened at a single US center
Groups:
- RUT058-60 vs Negative Control vs Positive Control: Each subject was their own control and received occlusive patches containing approximately 200 mg of all three (test article, negative control, and positive control) applied to abraded and non abraded skin sites in the scapular region of each subject's back.
Period: Overall Study
Arm/Group | RUT058-60 vs Negative Control vs Positive Control
Started | 43
Completed | 36
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Groups:
- RUT058-60 vs Negative and Positve Controls: All subjects who were enrolled, remained compliant and participated in all scheduled visits and received all study material applications were analyzed.
Arm/Group | RUT058-60 vs Negative and Positve Controls
Number analyzed (Participants) | 43
Age, Continuous [Median (Standard Deviation); unit: years] | 35 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  Latino | 2
  White | 37
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Irritation Score of RUT058-60 Hypochlorous Acid Solution (106 mg/L) on Healthy Human Skin
Description: Primary Analysis After a 23-hour ± 1-hour period of exposure, patches were removed, and the sites evaluated and visually scored for irritancy. The procedures will be repeated on the same test sites an additional twenty times. On each day,mean values, sample sizes, ranges, etc., of the irritation scores, for a total of six configurations, were recorded.
  Grading Scale for Visual Evaluation of Skin Condition: 0= no evidence of irritation, 1= minimal erythema, barely perceptible, 2= definite erythema, readily visible; minimal edema or minimal papular response, 3= erythema and papules, 4= definite edema, 5= erythema, edema, and papules, 6=' vesicular eruption, 7= strong reaction spreading beyond test site Visual observations of 3, 4, or 5 resulted in discontinuance of product application to that site. Observations of 6 or 7 were considered an adverse event and subject discontinued from the study.
Time Frame: 21 days
Population: Each subject had each study material (test, positive and negative controls) applied to separate abraded and non-abraded skin sites
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hypochlorous Acid Solution 106 mg/L-Abraded: 0.02 mL of the Test Product RUT058-60 applied to abraded skin sites.
- Sodium Lauryl Sulfate (0.1%) -Abraded: 0.02 mL of the Positive Control applied to abraded skin sites.
- Physiological Saline (0.9%), USP-Abraded: 0.02 mL of the Negative Control applied to abraded skin sites.
- Hypochlorous Acid Solution 106 mg/L- Non-Abraded: 0.02 mL of the Test Product RUT058-60 applied to non-abraded skin sites.
- Sodium Lauryl Sulfate (0.1%)- Non-Abraded: 0.02 mL of the Positive Control applied to non-abraded skin sites.
- Physiological Saline (0.9%), USP- Non-Abraded: 0.02 mL of the Negative Control applied to non-abraded skin sites.
Arm/Group | Hypochlorous Acid Solution 106 mg/L-Abraded | Sodium Lauryl Sulfate (0.1%) -Abraded | Physiological Saline (0.9%), USP-Abraded | Hypochlorous Acid Solution 106 mg/L- Non-Abraded | Sodium Lauryl Sulfate (0.1%)- Non-Abraded | Physiological Saline (0.9%), USP- Non-Abraded
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 36 | 36
units on a scale | 1.00 (0.68) | 2.46 (0.55) | 1.34 (0.44) | 0.58 (0.33) | 1.84 (0.58) | 0.82 (0.51)

ADVERSE EVENTS:
Arm/Group | RUT058-60 vs Negative and Positve Controls
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 5/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RUT058-60 vs Negative and Positve Controls (N=43)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Results from 36 subjects receiving all applications and completing all visits

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure Agreement